CLINICAL TRIAL: NCT05450744
Title: A Phase 1 Safety and Dose Finding Study of 131I -TLX101 Plus Standard of Care in Patients With Newly Diagnosed Glioblastoma
Brief Title: 131I-TLX-101 for Treatment of Newly Diagnosed Glioblastoma (IPAX-2)
Acronym: IPAX-2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 131I-TLX-101-002 (IPAX-2)
Record Dates: First submitted 2022-04-22; First posted 2022-07-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neoplastic Disease; Glioblastoma; Glioblastoma Multiforme
Keywords: Glioblastoma
MeSH Terms: conditions — Neoplasms; Glioblastoma | interventions — (18F)fluoroethyltyrosine

STUDY DESIGN:
Intervention Model Description: 3+3 ascending dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 131I-TLX101 + standard of care (Experimental)
  Interventions: Drug: 131I-IPA

INTERVENTIONS:
Drug: 131I-IPA — 131I-IPA: injection/solution administrated intravenously via infusion in ascending doses 18F-FET: injection/solution administrated intravenously
  Other Names: 18F-FET

SUMMARY:
This is an open label, single arm, parallel-group, multicentre, and dose finding study to evaluate the safety of ascending radioactive dose levels of 131I-TLX101 administered intravenously in combination with best standard of care in newly diagnosed GBM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form prior to any study related procedure and/or assessments being conducted.
2. Are Male or Female, and aged 18 years or older, at the time of signing the informed consent.
3. Have histologically confirmed intracranial glioblastoma (per WHO 2021 definition) following surgical resection. Tumours primarily localised in the infratentorial compartment will be excluded.
4. Have had prior surgery for glioblastoma, but no systemic therapy or radiation therapy for GBM.
5. Have a Karnofsky Performance Status ≥70.
6. Plan to begin chemoradiation therapy 3-6 weeks after surgical resection with Stupp regimen.
7. Have adequate organ function at Screening:

   7.1 Bone marrow: 7.1.1 Leukocytes ≥3,000/mL 7.1.2 Absolute neutrophil count ≥1500/mL 7.1.3 Platelets ≥100,000/mL 7.1.4 Haemoglobin ≥9g/dL 7.2 Liver function: 7.2.1 Total bilirubin ≤1.5×the upper limit of normal (ULN). For patients with known Gilbert's Syndrome ≤3×ULN is permitted 7.2.2 Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5×ULN 7.3 Renal function: 7.3.1 Serum/plasma creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min
8. Have at least 6 slides without staining or a tissue block (frozen or paraffin-embedded) available from a previous biopsy or surgery (tumour sample previously archived).
9. Have the capacity to understand the study and be able and willing to comply with all protocol requirements, including compliance with the radiation protection guidelines (including hospital admissions and isolation) that are applied by the treating institution to protect their contacts and the public.
10. Agree to practice adequate precautions to prevent pregnancy to avoid potential problems associated with radiation exposure to the unborn child.
11. Females must have a negative pregnancy test at screening and on dosing day, must not be lactating.

Exclusion Criteria:

1. Are unable to provide signed informed consent
2. Have had prior treatment for glioma, excluding surgery.
3. Are unable to undergo contrast-enhanced MRI.
4. Intend to be treated with tumor-treating fields prior to progression.
5. Have a history or evidence of delayed-type hypersensitivity (DTH)-dependent chronic infection (e.g., tuberculosis, systemic fungal or parasitic infection), potentially exacerbating under systemic corticoid therapy.
6. Have a known history of allergy TMZ, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
7. Have haemostaseologic conditions, precluding catheterisation or invasive procedures.
8. Have had phenylketonuria diagnosis previously
9. Have any medical condition that in the opinion of the Investigator may interfere with the participant's ability to adhere to the study or may impose a risk to the participant's health.
10. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 3 weeks of administration of study treatment except surgery on primary tumour.
11. Pregnant, breastfeeding or planning to get pregnant during the duration of the study.
12. Requirement of chronic administration of high dose corticosteroids or other immunosuppressant drugs. Limited or occasional use of corticosteroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
13. Have presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the participant at undue risk or unable to comply with study requirements. HIV-positive participants may be included in the study if they are on a stable dose of anti-retroviral therapy.
14. Have concurrent malignancies unless the patient has been disease-free without intervention for at least 2 years.
15. Have taken growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
16. Have serious, non-healing wound, ulcer, or bone fracture.
17. Have a requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
18. Have received any other IMP within 90 days prior to the planned administration of study drug.
19. Have uncontrolled Hashimoto's or Grave's disease
20. Have on-going and unresolved Grade ≥ 1 AEs following surgical resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and the grade (severity) of DLTs | 8 weeks from the first dose of IMP until discharge from the second dosem, up to 62 weeks.
  Incidence rate and the grade (severity) of DLTs based on the occurrence of Adverse Events (AEs) reported according to the NCI CTCAE v6.0. DLTs include any grade ≥ 3 events considered possibly related to the study drug, but excludes cerebral oedema, and haematological toxicity.
Safety, tolerability and RP2D | From screening until end of study, assessed over 62 weeks. TEAEs - units are frequency (percentage) and severity. Laboratory - safety laboratory including liver functions test, report mean and out of range.
  Assessing TEAEs type according to MedDRA (Medical Dictionary for Regulatory Activities), frequency, severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V5.0, seriousness, and relationship of study treatment will be assessed. Laboratory abnormalities will be assessed according to the NCI CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (4):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Olivia Newton John Cancer Research Institute/Austin Health, Melbourne, Victoria
- Institut für Nuklearmedizin und Endokrinologie, Linz, Austria
- UNMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No